CLINICAL TRIAL: NCT06625957
Title: A Randomized, Open-labeled, Multi-center, Active-controlled, Parallel-group Phase 3 Clinical Trial to Evaluate the Safety and Efficacy of NTCB02-1 Versus NTCB-C in Patients Who Require Parenteral Nutrition
Brief Title: Clinical Trial to Evaluate the Safety and Efficacy of NTCB02-1 in Patients Who Require Parenteral Nutrition
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NTCB02-301
Record Dates: First submitted 2024-10-02; First posted 2024-10-03 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Parenteral Nutrition
MeSH Terms: conditions — Hyperphagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NTCB02-1 (Experimental)
  Interventions: Drug: NTCB02-1
- NTCB-C (Active Comparator)
  Interventions: Drug: NTCB-C

INTERVENTIONS:
Drug: NTCB02-1 — 3 Days infusion
  Arms: NTCB02-1
Drug: NTCB-C — 3 Days infusion
  Arms: NTCB-C

SUMMARY:
A Randomized, Open-labeled, Multi-center, Active-controlled, Parallel-group Phase 3 Clinical Trial to Evaluate the Safety and Efficacy of NTCB02-1 versus NTCB-C in patients who require parenteral nutrition

ELIGIBILITY:
Inclusion Criteria:

* Those who are 19 years old or older at the screening visit
* Patients are expected to require PN for more than 3 days
* Patients who voluntarily signed the consent form

Exclusion Criteria:

* Patients are expected difficult to survive more than 3 days
* Patients BMI is over 30 kg/m2
* Patients having hypersensitivity to any peanut-, fish-, soy-, egg protein, or investigational drug
* Patients with difficult central venous line
* Patients judged to be unsuitable for this trial by investigators

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2025-07-18 (Estimated); Study Completion 2025-07-18 (Estimated)

PRIMARY OUTCOMES:
Occurance rate of adverse drug reaction | Day 1 to day 4

CONTACTS AND LOCATIONS:
Locations (5):
- South Korea (5):
  - National Cancer Center, Gyeonggi-do, Goyang-si
  - Chonnam National University Hwasun Hospital, Jeollanam-do, Hwasun-gun
  - Jeonbuk National University Hospital, Jeollabuk-do, Jeonju-si
  - Severance Hospital, Seoul, Seodaemun-gu
  - Seoul National University Bundang, Gyeonggi-do, Seongnam-si

IPD SHARING:
Plan to Share IPD: No